CLINICAL TRIAL: NCT02664714
Title: The Effects of Individual Pelvic Floor Muscle Training Versus Individual Treatment With Progression to Group Versus Group Training for Women With Stress Urinary Incontinence: Protocol for a Randomized Controlled Trial
Brief Title: Individual Pelvic Floor Muscle Training Versus Individual With Group Versus Group for Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Vilena Figueiredo Xavier, Director of Clinical Research, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5015537
Record Dates: First submitted 2015-12-16; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Incontinence Stress
Keywords: physiotherapy, perineometer, adherence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PFMT Individualized (Active Comparator): 12 Individualized pelvic floor muscle training:FAST CONTRACTIONS(repetitions) weeks 1(5x),2(10x),3(15x), 4(20x),5(30x),6(40x) 7-12(50x)SUSTAINED CONTRACTIONSNumber of series:weeks: 1 and 2(2), 3-6(3), 7-12(4)Repetitions:week 1(6) week 2(8), weeks 3-12 (10)Sustained contraction time/Resting time: weeks 1(2s/4s),2(3s/6s), 3(4s/8s) 4(5s/10s), 5(5s/5s), 6(5s/5s), 7(6s/6s),8(6s/6s), 9(8s/8s) 10(8s/8s), 11(10s/10s),12(10s/10s)
  Interventions: Other: PFMT
- PFMT individualized with group (Experimental): 12 Individualized pelvic floor muscle training:FAST CONTRACTIONS(repetitions) weeks 1(5x),2(10x),3(15x), 4(20x),5(30x),6(40x) 7-12(50x)SUSTAINED CONTRACTIONSNumber of series:weeks: 1 and 2(2), 3-6(3), 7-12(4)Repetitions:week 1(6) week 2(8), weeks 3-12 (10)Sustained contraction time/Resting time: weeks 1(2s/4s),2(3s/6s), 3(4s/8s)
  Interventions: Other: PFMT
- 12 group PFMT (Active Comparator): 12 Individualized pelvic floor muscle training:FAST CONTRACTIONS(repetitions) weeks 1(5x),2(10x),3(15x), 4(20x),5(30x),6(40x) 7-12(50x)SUSTAINED CONTRACTIONSNumber of series:weeks: 1 and 2(2), 3-6(3), 7-12(4)Repetitions:week 1(6) week 2(8), weeks 3-12 (10)Sustained contraction time/Resting time: weeks 1(2s/4s),2(3s/6s), 3(4s/8s)
  Interventions: Other: PFMT

INTERVENTIONS:
Other: PFMT — Participating volunteers of all groups will receive guidance about the anatomy and function of the pelvic floor muscles (PFM) and how to perform a properly contraction: as strong as possible and eliminating at the most the contraction of the gluteus, abdominals and adductors. For all groups it will be used the same protocol which was developed for this study, with progression parameters of the PFMT based on the recommendations for the strength training of the American College of Sports Medicine (VICKI, 2001).
  Other Names: pelvic floor muscles training

SUMMARY:
The aim of this study is to evaluate if the training of pelvic floor muscles, which associates an individualized treatment progressing to a group treatment, would be more effective than an individualized training only or groups only.

Methods: Randomized controlled study which will be done from January to December of 2016, on Laboratory of Women's Health Research, Federal University of São Carlos-SP, Brazil.

Inclusion criteria: women with stress UI, older than 18 years old. The sample size calculation was performed using the GPower Software (3.1.5, Germany) and it was estimated a sample of 30 women in each group. The volunteers will be assessed before the intervention by a urinary symptoms evaluation form, King's Health Questionnaire, miccional diary, PERFECT scheme and perineometry.

After the evaluation will be performed the randomization of the volunteers by a blinded investigator and the volunteers will be allocated into three groups:

Group 1: Individualized Training Group 2: Individualized training with progression to group training Group 3: Group training only

For all groups it will be used the same protocol that was prepared according to the recommendations of the American College of Sports Medicine. Later, volunteers will be reassessed after 12 treatments, three months and six months (from the discharge date). It will be added in the reassessment the Self-efficacy Scale for Pelvic Floor Exercises Practice.

Primary outcome: severity measures of the King's Health Questionnaire.

Secondary outcome: miccional diary, PERFECT scheme, perineometry and Self-efficacy scale for Pelvic Floor Exercises Practice. Data normality will be tested by the Shapiro-Wilk test (SPSS 19.0). The comparison between the evaluations will be performed by ANOVA, and the comparison between groups will be performed by Student t-test (independent measures). In order to measure the practical significance of the data, the effect size and the confidence interval (CI) will be calculated. A 5% significance level will be assumed. This study was approved by the Research Ethics Committee of the Federal University of São Carlos, São Carlos- SP, Brazil (Protocol 1207393).

DETAILED DESCRIPTION:
This is a blinded randomized controlled clinical trial. Data collection will be performed at the Women's Health research laboratory (WHRL), allocated in the Department of Physical Therapy of Federal University of São Carlos, from January 2016 to December 2016.

The project was approved by the Research Ethics Committee (REC) of Federal University of São Carlos (UFSCar) (Number 1207393). Patients will receive information about the research and those who consent to participate, will sign the free informed consent form.

The sample size calculation was performed using the GPower Software (3.1.5, Germany) based on the study of Pereira et al (2011) considering the intergroup comparison of data post treatment of the severity measurement of the King's Health Questionnaire. It was considered the ANOVA (repeated measures), 80% power, effect size of 0.40 and 5% of significance level, being estimated a sample size of 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* women from the age of 18 years old who present urinary incontinence stress

Exclusion Criteria:

* urge urinary incontinence (UUI) in an isolated form, neuromuscular diseases, other diseases (asthma, tumors, heart failure, absence of pelvic floor muscle contraction (grade 0) verified by modified Oxford scale, urinary infection, difficulty in understanding the study procedures, uncontrolled hypertension, presence of severe prolapse (visible prolapse in the vaginal opening), women with UI who have done physical therapy in the last 12 months, pregnancy,puerperium.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
severity measures of the King's Health Questionnaire | 6 months
  In the first assessment volunteers will answer the King's Health Questionnaire

SECONDARY OUTCOMES:
mictional diary, PERFECT scheme, perineometry and Self-efficacy scale for Pelvic Floor Exercises Practice | 6 months
  the volunteer will be placed in the supine position with flexed hip and knees. Initially, it will be observed the vaginal mucosa condition, the presence of atrophies, sensitivity, pelvic organ prolapse and the tone of the vaginal wall. Then, it will be performed the muscle function evaluation through the PERFECT scale which was developed, the researcher will introduce the index finger about 4 cm into the volunteer vaginal canal and will guide her to contract the PFM.After, it will be evaluated the pelvic floor muscles contraction pressure through the Peritron equipment (Cardio Design,Australia) and is equipped with a vaginal probe. The perineometer probe will be coated with a male non-lubricated condom and will be introduced with KY® lubricant gel into the volunteer's vagina.

CONTACTS AND LOCATIONS:
Overall Officials: Vilena F Xavier, Principal Investigator — Programa de Pós-Graduação em Fisioterapia - UFSCar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BØ K, LARSEN S, OSEID S, et al. Knowledge about and ability to correct pelvic floor muscle exercises in women with urinary stress incontinence. Neurourol Urodyn. 1988;7:261-262. BØ K, TALSETH T, VINSNES A: Randomized controlled trial on the effect of pelvic floor muscle training on the quality of life and sexual problems in genuine stress incontinent women. Acta Obstet Gynecol Scand, 79:598-603, 2000. BO K, SHERBURN M. Evaluation of female pelvic-floor muscle function and strength. Phys Ther; 85 (3): 269 -82, 2005. BØ, K. AND HILDE, G. Does it work in the long term?-A systematic review on pelvic floor muscle training for female stress urinary incontinence. Neurourol. Urodyn., 32: 215-223, 2013. BORELLO-FRANCE DF, ZYCZYNSKI HM, DOWNEY PA, RAUSE CR, WISLER JA. Effect of pelvic floor muscles exercise position on continence and quality of life outcomes in women with stress urinary incontinence.Phys Ther. 86:974-86, 2006.
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- See also: test link — http://www.ppgft.ufscar.br/